CLINICAL TRIAL: NCT07380126
Title: The Effect of Functional Crown Lengthening Versus Deep Margin Elevation on Periodontal Tissues (A Randomized Clinical Trial With Biochemical Analysis)
Brief Title: The Effect of Functional Crown Lengthening Versus Deep Margin Elevation on Periodontal Tissues
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-Rec IM022410
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: TNF Alpha
Keywords: Functional Crown lengthening; Deep Margin Elevation; TNF-α

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional crown lengthening (Experimental): patients will undergo functional crown lengthening by raising a full thickness flap with osseous resection to establish a distance of 3 mm between the cervical margin of the cavity and the bone crest. Osteoplasty was performed in the adjacent and neighboring tooth surfaces to accomplish a smooth bone contour. The flaps will then be sutured in their new position
  Interventions: Procedure: Functional Crown lengthening
- Deep Margin Elevation (Active Comparator): patients will undergo deep margin elevation through a two-step direct restoration performed using the concepts of Progressive Matrixing and Wedging where the Deep subgingival cavity margin will be acquired. Then isolation by rubber dam. A curved matrix will seal the margin without any gingival or rubber dam entrapped in between. One step adhesive system will be performed under rubber dam isolation. Composite resin base is applied to raise the margin by about 2 mm. A bulk fill packable or flowable composite can be used. Finishing will be done using polishing strips and disks. Finally a bitewing radiograph will be taken to check the presence of overhangs or gaps before the final restoration.
  Interventions: Procedure: Deep Margin Elevation

INTERVENTIONS:
Procedure: Functional Crown lengthening — patients will undergo functional crown lengthening by raising a full thickness flap with osseous resection to establish a distance of 3 mm between the cervical margin of the cavity and the bone crest. Osteoplasty was performed in the adjacent and neighboring tooth surfaces to accomplish a smooth bone contour. The flaps will then be sutured in their new position
  Arms: Functional crown lengthening
Procedure: Deep Margin Elevation — patients will undergo deep margin elevation through a two-step direct restoration performed using the concepts of Progressive Matrixing and Wedging where the Deep subgingival cavity margin will be acquired. Then isolation by rubber dam. A curved matrix will seal the margin without any gingival or rubber dam entrapped in between. One step adhesive system will be performed under rubber dam isolation. Composite resin base is applied to raise the margin by about 2 mm. A bulk fill packable or flowable composite can be used. Finishing will be done using polishing strips and disks. Finally a bitewing radiograph will be taken to check the presence of overhangs or gaps before the final restoration.
  Arms: Deep Margin Elevation

SUMMARY:
The present study will evaluate and compare the effect of functional CL and DME in the treatment of posterior teeth with class II caries clinically and on the level of TNF-α in the GCF of treated teeth.

Clinical evaluation of periodontal tissue in the form of probing depth as a primary outcome, clinical attachment level, plaque index, bleeding index, gingival index, pink aesthetic score, Radiographic evaluation of biological width and the level of TNF-α in the GCF as a secondary outcome.

DETAILED DESCRIPTION:
In dental practice, restoring cavitated proximal caries lesions is a common routine procedure in dental clinics. However, subgingival margins reaching below the cementoenamel junction are known to have a common clinical concern, especially when restoring severely destructed Class II caries. Ideally, the correct choice of treatment plan is critical to ensure successful outcomes (Padbury et al., 2003).

The use of direct adhesive restoration to restore large interproximal defects is not an ideal treatment option. Due to their size, such defects usually require indirect adhesive restorations. However, this appears to be challenging since cavity preparation, impression taking, the adhesive-bonding procedure, and proper moisture control may be impeded. These challenges are usually overcomed by functional crown lengthening (Mangani et al.,2015; Juloski et al.,2018).

Functional Crown lengthening is a surgical procedure to expose the gingival margins by apical displacement of the supporting periodontal structures, thus can facilitate an access and adequate isolation to achieve the optimum position of deep restorations and avoid violating the biological width (Magne & Spreafico, 2012; Sarfati & Tirlet, 2018).

The biological width is defined as the gingival attachment along the root surface, from the most coronal portion of the epithelium attachment to the most apical portion of the connective tissue attachment (Gargiulo et al.,1961). Therefore, a recommended distance of 3 mm or more between the restorative margins and the alveolar crest is considered necessary to avoid detrimental effects on neighbouring soft and hard periodontal tissues (Ingber et al.,1977; Lanning et al., 2003). The violation of the biological width results in severe gingival inflammation and consequently deep pocket formation or gingival recession, in addition to bone level reduction (Nugala et al., 2012).

Recurrence usually occurs particularly in patients with thick biotypes or when surgery comprises only gingivectomy. Moreover, recurrence leads to restoration limits being replaced sub-gingivally, whereas surgery aims to place them sub-gingivally (Ganji et al.,2012)..

A more conservative approach is the deep marginal elevation (DME), which is considered an atraumatic procedure advocated in the presence of deep cervical margins (Dietschi & Spreafico,1998; Veneziani,2010).

The concept of "deep margin relocation" was introduced in 1998 by Dietschi and Spreaficoas a new approach to deep caries. It was later renamed "deep margin elevation" by Magne and Spreafico in 2012. It is a procedure done to raise the margins of the tooth to either an equi-gingival or supra-gingival position using restorative materials. This technique is referred to by different names, including the "open sandwich technique," "proximal box elevation," and the "margin elevation technique" (Dietschi & Spreafico,1998; Dietschi et al.,2003).

A dry working field is crucial to the success of restoration, especially in deep cavities reaching the Cemento-enamel junction. The presence of saliva and blood causes contamination and deterioration to the restoration and affects the bonding to the tooth structure (Keys & Carson,2017).

DME allows appropriate placement of a rubber dam to a perfectly placed margin, adequate light-curing depth to the margin of restoration, accessibility to proper oral hygiene, and an ultraconservative approach to evaluate bone and soft tissue (Frankenberger et al.,2013; Zaruba et al.,2013). Studies have shown promising results using DME and high survival rates of up to 90% over a 12-year clinical evaluation (Bresser et al.,2019).

A randomized clinical trial compared the clinical results of crown lengthening and DME in posterior teeth. At 180 days, clinical attachment loss was higher in the surgical group (Bresser et al., 2019). Many studies have reported that DME procedures do not negatively affect periodontal health status and suggest they are well tolerated by the periodontium when proper isolation is achieved (Frese et al.,2014; Sarfati & Tirlet, 2018).

However, the gingival phenotype must be analysed as among teeth treated with subgingival restorations, those presenting <2 mm of keratinized tissue showed higher gingival index (Stetler & Bissada,1987).

Debate continues as to whether a non-invasive elevated margin technique or surgical CL is the better strategy for facilitating the placement of large direct composite resin restorations. Though a conservative approach is often advocated, it fails in situations that demand change in the shape of tissues around the tooth for restoration (Sarfati & Tirlet, 2018).

To the best of our knowledge, no previous study measured the effect of crown lengthening on inflammatory biomarkers in the gingival crevicular fluid in comparison to deep margin elevation in posterior teeth with deeply located proximal margins.

ELIGIBILITY:
Inclusion Criteria :

1. Patients aged 20-50 years
2. Both genders
3. Patients free from any systemic disease that may affect the treatment (Greenberg & Glick, 2012)
4. Patients with intact periodontium
5. Patients are ready to comply with oral hygiene measures.
6. Patients having Posterior teeth with carious cavities and/ or restorations in need of replacement on proximal surfaces, where the cervical margin of the cavity is at a distance less than 3 mm to the bone crest (Cyana et al.,2013).
7. Patients with thick phenotype having gingival thickness > 1mm (Aimetti et al,2008).
8. Patients with keratinized tissue width ≥ 2mm

Exclusion criteria:

1. Pregnant and lactating females
2. Smokers
3. Drug abusers.
4. Patients with persistent poor oral hygiene
5. Patients with proximal margins beyond the bone level
6. Patients with developmental dental anomalies
7. Patients undergoing or will start orthodontic treatment

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Probing depth | Clinical measurements preoperative and will be repeated at 1, 3, and 6 months
  Will be measured from the gingival margin to the depth of the pocket at four points (mesio-facial, mid-facial, disto-facial and mid-lingual) to the nearest millimeter using UNC-15 periodontal probe. The average of the three facial points will be recorded as the facial probing depth (FPD), while the mid-lingual point will be recorded as the lingual probing depth.

SECONDARY OUTCOMES:
Biochemical evaluation | Biochemical measurements preoperative and will be repeated at 1, 3 and 6 months
  GCF samples will be collected to measure the level of TNF-α in treated teeth. Before sampling, the adjacent teeth will be isolated with cotton rolls. Crevicular fluid will be collected on perio paper strips placed parallel to the long axis of the tooth of concern in the gingival sulcus until mild resistance is felt and kept for 30 seconds and pooled in reduced transport fluid (RTF) medium for biochemical analysis. GCF collected samples contaminated with blood and saliva will be discarded

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A. Khattab, Associate Professor, Study Director — Faculty of Dentistry - Ain shams university

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Padbury A Jr, Eber R, Wang HL. Interactions between the gingiva and the margin of restorations. J Clin Periodontol. 2003 May;30(5):379-85. doi: 10.1034/j.1600-051x.2003.01277.x. PMID 12716328
- [Background] Aimetti M, Massei G, Morra M, Cardesi E, Romano F. Correlation between gingival phenotype and Schneiderian membrane thickness. Int J Oral Maxillofac Implants. 2008 Nov-Dec;23(6):1128-32. PMID 19216284